CLINICAL TRIAL: NCT06083558
Title: Pain and Nausea in the Post-anesthesia Care Unit Following Gallbladder Surgery - a Registry Study Using National Data From Gallriks and the Swedish Perioperative Register (SPOR)
Brief Title: Pain and Nausea After Gallbladder Surgery
Status: Recruiting | Type: Observational
Sponsor: Umeå University (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: GALLSPOR
Record Dates: First submitted 2023-10-05; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: PONV; Postoperative Pain; Postoperative Complications; Gall Bladder Disease
Keywords: cholecystectomy
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Pain, Postoperative; Postoperative Complications; Gallbladder Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is primarily an exploratory study of quality registry data for a swedish national cohort of patients who have undergone gallbladder surgery or ERCP, with the aim of investigating the occurrence of pain and PONV (Postoperative Nausea and Vomiting) after gallbladder surgery. Furthermore, the investigators will explorer if there are factors related to the patient or the surgical procedure that are associated with a higher risk of PONV or pain.

DETAILED DESCRIPTION:
The project is a registry study with linked data from the Swedish national registry for gallbladder surgery (Gallriks) and the Swedish Perioperative Register (SPOR).

In SPOR, multiple variables are recorded and the main categories include patient characteristics, process data (e.g., times, operating room, planning, cancellations), surgical data (diagnosis, procedure, anesthesia type, times, deviations), and postoperative data (e.g., pain, nausea, complications, times, postoperative care level). The main variables of interest in this project are postoperative nausea and vomiting (PONV) and pain. In SPOR, it is possible to register whether the patient experienced nausea or vomiting and to assess pain in the immediate postoperative period during the stay at the postoperative recovery unit (PACU). The mean time of stay at PACU after gallbladder surgery in Sweden is 3.5 hours.

Gallriks records data related to gallstone surgery, including preoperative factors (including patient's illness), surgical processes, and postoperative outcomes up to 6 months after surgery.

The investigators have estimated that it is possible to include at least 50% of all gallstone surgeries in Sweden, which corresponds to a range of 7,000-8,000 patients per year.

Both quality registers are housed at the Uppsala Clinical Research Center (UCR), which will perform the data linkage. The data extraction process will start with the surgical cases in Gallriks and match them with SPOR. The database delivered to the research group will contain only pseudonymized personal data, with personal identification numbers and names removed.

The objectives of the study are:

* Describe the risk of early PONV (Postoperative Nausea and Vomiting) and pain during the PACU stay following gallstone surgery.
* Identify factors associated with early PONV and pain.
* Test the hypothesis that total intravenous anesthesia has a lower risk of PONV and pain at the PACU compared to inhalation-based anesthesia.
* Test the hypothesis that the addition of a regional block reduces the risk of PONV and pain during the PACU stay.
* Test the hypothesis that patients who experience PONV and/or pain in the postoperative ward have a higher risk of postoperative complications up to 6 months after surgery.

The primary outcome measures are:

* Risk of PONV in the postoperative ward (number of surgical cases with nausea and/or vomiting) / [total number of surgical cases].
* Median pain score (NRS) in the postoperative ward.
* Risk of severe pain (NRS>=7) [number of surgical cases with NRS>=7] / [total number of surgical cases].
* Percentage of patients with complications, unplanned hospitalizations, or reoperations after 30 days and 6 months.
* Based on the data in SPOR and Gallriks, identify factors associated with the primary outcome measures. Variables hypothesized to be associated include gender, age, illness, preoperative pain, type of anesthesia, type of surgery, and length of hospital stay.
* Specifically examine whether total intravenous anesthesia or regional blockade reduces the risk of PONV/pain and whether PONV/pain increases the risk of postoperative complications.

The data will be described using descriptive methods, and associations will be analyzed through univariate and multivariate analysis.

The study database is planned to include the procedures performed during the years 2016-2025. Databases will be delivered on a yearly basis. Analysis and reports/manuscripts from the study might include parts of the whole study period of 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Primary gallstone surgery
* Adult patients (>=18 years)
* Procedure performed between 2016 and 2025
* Surgical procedure registered in the national quality registry Gallriks.

Exclusion Criteria:

* If multiple surgeries on the same patient in the study database, subsequent procedures to the first procedure is excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients that had undergone gallbladder surgery in Sweden.
Sampling Method: Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting | Through the stay at the PACU, an average of 3.5 hours
  Incidence of PONV in the postoperative ward (number of surgical cases with nausea and/or vomiting) / [total number of surgical cases].
Postoperative Pain | Through the stay at the PACU, an average of 3.5 hours
  Median pain score (NRS) in the postoperative ward.
  NRS = Numerical Rating Scale 0-10. 0 = No pain and 10 = Worst imaginable pain
Severe postoperative pain | Through the stay at the PACU, an average of 3.5 hours
  Incidence of severe pain (NRS>=7) [number of surgical cases with NRS>=7] / [total number of surgical cases].
  NRS = Numerical Rating Scale 0-10. 0 = No pain and 10 = Worst imaginable pain
Complications after surgery | up to 6 month
  Percentage of patients with complications, unplanned hospitalizations, or reoperations after 30 days and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Wallden, MD PhD, Principal Investigator — Umeå University
Locations (1):
- Umeå University, Dept of surgical and perioperative sciences, Sundsvall, X, Sweden